CLINICAL TRIAL: NCT02041130
Title: Renal Sympathectomy in Heart Failure (the RESPECT-HF Study) - a Study of Renal Denervation for Heart Failure With Preserved Ejection Fraction
Brief Title: Renal Denervation in Heart Failure Patients With Preserved Ejection Fraction (RESPECT-HF)
Acronym: RESPECT-HF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: University of Otago (Other); Wellington Hospital (Other Government); University of Auckland, New Zealand (Other); Monash University (Other); Tan Tock Seng Hospital (Other); Changi General Hospital (Other); Singapore Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSRB: 2013/00457
Record Dates: First submitted 2013-10-28; First posted 2014-01-20 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Heart Failure
Keywords: Heart Failure; Heart Failure with Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal Denervation and standard medical management (Experimental): Renal Denervation (RDN) is a simple catheter procedure removing excess nerve signals to and from the kidneys. The renal denervation system consists of a small steerable treatment catheter and an automatically-controlled treatment delivery generator.
  A guiding catheter is inserted through a tiny incision in the groin into the femoral artery to direct the treatment catheter to the renal arteries. The treatment catheter delivers high -frequency radio waves, called radiofrequency wavees, to 4-6 locations within each of the two renal arteries. the energy delivered is about 8 watts and aims to disrupt the nerves and lower blood pressure over a period of months. The procedure takes 40-60 minutes.
  Interventions: Device: Renal Denervation
- Contorl and Standard Medical Management (No Intervention): Continued medical management will comprise management of all cardiovascular risk factors (hypertension, diabetes, dyslipidaemia) in accord with international guidelines. Lifestyle and dietary counselling will also be part of the patient management. As there is no established evidence-based pharmacotherapy for HFPEF per se, therapy aimed at HF specifically will adopt treatments recommended for HFREF with prescription of diuretic, ACE inhibitor/ARB, beta blocker and mineralocorticoid antagonist accordingly.

INTERVENTIONS:
Device: Renal Denervation
  Other Names: Symplicity Catheter System; renal sympathetic denervation; renal ablation
  Arms: Renal Denervation and standard medical management

SUMMARY:
Investigators will test a new approach to a form of heart failure (HF) with no current treatment proven to reduce death rates or hospitalisations. Over a third of HF cases have preserved ejection fraction (HFPEF) often on a background of high blood pressure (BP). These "stiff" hearts pump strongly but fill inefficiently resulting in poor exercise capacity and high death rates. Treatments that help when heart pumping action is poor are of no benefit in HFPEF. Recently a simple catheter procedure removing excess nerve signals to and from the kidneys ("renal denervation"; RDN) has been able to reduce BP in patients with high BP resistant to multi-drug treatment. Through removing excess nervous drive to the kidneys, heart and circulation this treatment has promise in HF. The investigators will compare effects of RDN and standard medical treatment on heart function, exercise capacity and quality of life in 144 patients with HFPEF

DETAILED DESCRIPTION:
Rationale for Research:- Heart failure (HF) is common and lethal. It is the most common diagnosis for medical admissions over 60 years of age, carries a >50% 5 year mortality and accounts for 1-2% of the total national health care budget. HF with preserved ejection fraction (HFPEF) includes over a third of HF cases presenting to New Zealand and Singapore Hospitals and has no treatment proven to reduce mortality or recurrent admissions. Renal denervation (RDN) has proven efficacy in refractory hypertension and its array of effects upon haemodynamic status, neurohumoral activity and renal function make it a rational candidate therapy in HFPEF.

Aims:- The investigators aim to conduct a phase 2 randomized controlled trial of RDN in HFPEF to determine effects upon cardiac structure and function, exercise capacity, and quality of life.

Primary Hypothesis: RDN will reduce left atrial volume index (LAVi) and/or left ventricular mass index (LVMi) on cardiac magnetic resonance imaging (cMRI).

Secondary Hypotheses: RDN will:

1. improve exercise capacity and functional status.
2. reduce E/e' and echocardiographic grade of diastolic dysfunction.
3. reduce circulating biomarkers of cardiac load, interstitial fibrosis and inflammation.
4. improve ventricular-vascular function.
5. improve Minnesota Living with Heart Failure (MLWHF) scores.
6. reduce the composite end-point of death or re-admission with HF.

Design and Methods:- Renal denervation will be tested as a therapy for HFPEF in a multi-centre open, randomized controlled trial of bilateral renal artery denervation compared with ongoing medical management. Sample size (n=144) will be sufficient to provide 90% power to detect clinically relevant effects on the primary endpoints of change in left atrial volume and left ventricular mass over 6 months post-RDN. Secondary end-points will include assessment of exercise capacity, ventricular-vascular coupling, biomarkers (of cardiac haemodynamic load, fibrosis, inflammation and cardiomyocyte loss), quality of life and cardiovascular events.

Research Impact:- Heart Failure with Preserved Ejection Fraction (HFPEF) is common, triggers recurrent hospital admissions has a high mortality and carries a high burden of health care costs. There is currently no treatment which reduces admissions or improves survival in this condition. If efficacy is proven, renal nerve denervation represents a simple, cost-effective, one time only, approach that will find rapid uptake potentially for thousands of cases.If the current proposal generates positive results (followed by positive phase 3 trials) the investigators conservatively estimate RDN may reduce both mortality and HF admissions in HFPEF by at least 30%.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HFPEF (based upon ESC diagnostic criteria9)

   1. Symptoms and signs of heart failure; NYHA Class II or higher
   2. Left ventricular ejection fraction 50% or greater on echocardiography
   3. Echocardiographic evidence of left ventricular diastolic dysfunction (echo-Doppler E/e' > 15 )AND/OR plasma NTproBNP > 220pg/ml.
2. Episode of acute decompensation (ADHF)
3. Patients with and without background hypertension may be recruited. In the case of patients with background hypertension (ie history of fulfilling the diagnostic WHO criteria for hypertension: SBP > 140 mmHg and/or DBP > 90 mmHg) those with both controlled (<140/90mmHg by 24 hour ambulatory BP) and inadequately controlled BP (on 3 anti-hypertensive drugs including a diuretic) can be recruited.

Exclusion Criteria:

1. Known secondary cause of hypertension
2. Renal artery stenosis >30% or anatomy otherwise unsuitable for RDN.
3. Heart failure with reduced LV ejection fraction (LVEF < 50%).
4. Estimated glomerular filtration rate (eGFR) of < 30mL/min/1.73m2 (MDRD calculation).
5. Systolic blood pressure < 105mmHg.
6. Implanted pacemaker, prosthetic heart valve or other precluding cMR scanning.
7. Medical condition adversely affecting safety and/or effectiveness of the participant (including peripheral vascular disease, abdominal aortic aneurysm, thrombocytopenia or atrial fibrillation).
8. Pregnant, nursing or planning to be pregnant.
9. Uncontrolled atrial fibrillation, ie with heart rate over 120 bpm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Compare the changes in left atrial volume index (LAVi) and/or left ventricular mass index (LVMi) on cardiac magnetic resonance imaging (cMRI) between baseline and 6 months | baseline, 6 months

SECONDARY OUTCOMES:
Compare the changes in exercise capacity and functional status as assessed by maximal oxygen consumption (VO2max) on cardiopulmonary exercise testing and by 6-minute walk test between baseline and 6 months | baseline, 6 months
Compare the changes in chocardiographic grade of diastolic dysfunction as assessed by Tissue Doppler E/e', (a non-invasive estimate of left atrial filling pressure). | baseline, 6 months
Compare the changes in biomarkers of cardiac load and interstitial fibrosis as assessed by plasma assays of relevant biomarkers | baseline, 6 months
  The biomarkers of cardiac load and interstitial fibrosis as assessed by plasma assays of markers of ventricular and atrial haemodynamic load, other neurohormones contributing to HF pathophysiology, cytokine markers of inflammation and remodelling, markers of cardiac fibrosis, a marker of cardiomyocyte loss.
Compare the changes in ventricular-vascular function as evaluated by echocardiographic measures of arterial elastance, Left Ventricular (LV) end-systolic elastance, LV filling pressure, and LV diastolic stiffness between baseline and 6 months | baseline, 6 months
Compare the changes of Quality of life as assessed by the Minnesota Living with Heart Failure between baseline and 6 months. | baseline, 6 months
Compare the difference in composite end-point of death or hospitalization with Heart Failure between control arm and treatment arm | baseline, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Mark Richards, MBChB, MD (Distinction), PhD, Study Chair — University of Otago, Christchurch; Henry Krum, MBBS, PhD, FRACP, FCSANZ, Principal Investigator — Monash University; Carolyn Lam Su Ping, MBBS, MRCP, MS, Principal Investigator — National University Heart Centre, Singapore
Locations (7):
- Monash University, Melbourne, Australia
- New Zealand (3):
  - The University of Auckland, Auckland
  - University of Otago, Christchurch
  - Wellington Hospital, Wellington
- Singapore (3):
  - Changi General Hospital, Singapore
  - National University Heart Centre, Singapore
  - Tan Tock Seng Hospital, Singapore